CLINICAL TRIAL: NCT05201300
Title: Comparison of Remimazolam and Propofol Anesthesia on Hemodynamic and Recovery Profile in Elderly Patients
Brief Title: Remimazolam and Propofol Anesthesia in Elderly Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, Jong Yeop Kim, Professor, Ajou University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: AJIRB-MED-INT-21-651
Record Dates: First submitted 2022-01-03; First posted 2022-01-21 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Hemodynamics
MeSH Terms: interventions — Propofol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Remimazolam 6 (Experimental): Remimazolam starts at 6 mg/kg/hr until loss of consciousness
  Interventions: Drug: Remimazolam Besylate 6 mg/kg/hr
- Remimazolam 12 (Experimental): Remimazolam starts at 12 mg/kg/hr until loss of consciousness
  Interventions: Drug: Remimazolam Besylate 12 mg/kg/hr
- Propofol (Active Comparator): Propofol starts at a target controlled infusion 4 µg/ml until loss of consciousness.
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Remimazolam Besylate 6 mg/kg/hr — Patients will receive remimazolam at 6 mg/kg/hr by continuous infusion until loss of consciousness.
  Other Names: Byfavo
  Arms: Remimazolam 6
Drug: Remimazolam Besylate 12 mg/kg/hr — Patients will receive remimazolam at 12 mg/kg/hr by continuous infusion until loss of consciousness.
  Other Names: Byfavo
  Arms: Remimazolam 12
Drug: Propofol — Patients will receive propofol at a target controlled infusion 4 µg/ml until loss of consciousness.
  Other Names: Fresofol
  Arms: Propofol

SUMMARY:
Remimazolam is a recently developed ultra-short agonist acting at the benzodiazepine binding site of the gamma-aminobutyric acid (GABA)A receptor. Remimazolam has a combination of the hemodynamic stability of benzodiazepines and the advantages of propofol, such as rapid onset, short duration of action, and improved controllability.

A recent study showed that the efficacy of two induction doses of remimazolam (6 and 12 mg/kg/h) as a sedative for general anesthesia was not inferior to propofol (2.0-2.5 mg/kg), and hemodynamically more stable. On the other hand, a study on the emergence time and quality between propofol and remimazolam showed inconsistent results.

The purpose of this study is to compare remimazolam to propofol on the intraoperative hemodynamic changes and recovery profiles, when used in combination with remifentanil in elderly patients undergoing general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* ASA I, II patients over 65 years old undergoing general anesthesia

Exclusion Criteria:

* cardiac surgery
* neurosurgery
* liver surgery
* uncontrolled hypertension
* bronchial asthma
* body mass index ≥ 30 kg/m2
* severe heart, liver, kidney disease

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 69 (Actual)
Dates: Start 2022-02-02 (Actual); Primary Completion 2022-11-25 (Actual); Study Completion 2023-01-18 (Actual)

PRIMARY OUTCOMES:
difference in the decreased mean arterial pressure | from the start of anesthetics (propofol or remimazolam) injection to the 5 minutes after extubation
  difference between baseline mean arterial pressure and lowest mean arterial pressure

CONTACTS AND LOCATIONS:
Locations (1):
- Ajou University Hospital, Suwon, Gyeonggi-do, South Korea